CLINICAL TRIAL: NCT06472063
Title: Upfront Surgery Versus NeoAdjuvant Chemotherapy Followed by Surgery for Resectable Advanced Gastric Cancer (SNAC Study): An Observational Retrospective Multicenter Study With Matched Treatment Comparison
Brief Title: Upfront Surgery Versus NeoAdjuvant Chemotherapy Followed by Surgery for Resectable Advanced Gastric Cancer: SNAC Study
Acronym: SNAC
Status: Recruiting | Type: Observational
Sponsor: San Luigi Gonzaga Hospital (Other)
Collaborators: Azienda Ospedaliera Universitaria Senese (Other); IRCCS Ospedale San Raffaele (Other); Federico II University (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Ospedaliero Universitaria Policlinico Modena (Other); Istituti Tumori Giovanni Paolo II (Network); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); ASST Grande Ospedale Metropolitano Niguarda (Other); Azienda Ospedaliera Sant'Anna (Other); Ospedale di Circolo - Fondazione Macchi (Other); Ospedale San Donato (Other); Government hospital in Forlì, Italy (Other); Istituti Ospitalieri di Cremona (Other); Azienda Ospedaliero-Universitaria Careggi (Other); Azienda ULSS di Verona e Provincia (Other); Azienda Ospedaliera di Perugia (Other); A.O. Ospedale Papa Giovanni XXIII (Other); Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Provincia Autonoma di Trento (Other Government); University of Florence (Other); Ospedale M. Bufalini Cesena (Other); Azienda Ospedaliera di Padova (Other); Ospedale Guglielmo da Saliceto, Piacenza (Unknown); Azienda Ospedaliera San Gerardo di Monza (Other); A.O.U. Città della Salute e della Scienza (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Ospedale Santo Stefano (Other); Policlinico Abano Terme (Other); Istituto Europeo di Oncologia (Other); Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other); Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Rossella Reddavid, MD, PhD, San Luigi Gonzaga Hospital
Other Study IDs: SNAC01
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer
Keywords: upfront surgery; perioperative treatment; D2 lymphadenectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Lead

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- upfront D2 gastrectomy (S): patients submitted to upfront D2 gastrectomy
- pre- or perioperative treatment and D2 gastrectomy (NAC): patients who underwent pre- or perioperative treatment and D2 gastrectomy
  Interventions: Other: pre- or perioperative treatment and D2 gastrectomy

INTERVENTIONS:
Other: pre- or perioperative treatment and D2 gastrectomy — pre- or perioperative treatment and D2 gastrectomy
  Other Names: perioperative treatment
  Groups: pre- or perioperative treatment and D2 gastrectomy (NAC)

SUMMARY:
Based on the concerns about the actual low strength of evidence of the efficacy of NAC on survival of proper gastric cancer treated with adequate D2 gastrectomy as compared to the results of optimal upfront surgery (S), and considering the actual difficulties of additional RCTs, the aim of this study is to assess the non-inferiority of upfront surgery alone with optimal D2 dissection compared to NAC regimens followed by surgery. Methods: This is a nationwide Multicenter observational retrospective study with matched comparison of two therapeutic strategies (NAC vs S). We will include patients with cT>2, every cN M0, or with every T and N+ M0, histologically proven adenocarcinoma of the stomach, submitted either to pre- or peri-operative treatment and D2 gastrectomy or to upfront D2 gastrectomy, between January 2012 and December 2019, followed by adjuvant treatment when recommended.

All patients matching the inclusion/exclusion criteria will be registered into the study and classified into one of the two arms: a, patients who underwent pre- or perioperative treatment and D2 gastrectomy (NAC) or b, patients submitted to upfront D2 gastrectomy (S). Given the results reported in the "FLOT" trial, a 3-years OS of 55% in the control arm (NAC) was assumed. Three-year OS in the experimental arm (S) was assumed to be 47.4% under the null hypothesis of inferiority and 55% under the alternative hypothesis of non-inferiority. A sample size of 684 patients (342 in each arm) achieves 80% power to detect a non-inferiority margin Hazard Ratio of 1.25

ELIGIBILITY:
Inclusion Criteria:

* 3.1.1. Locally advanced (T>2 any N or N+ any T) histologically proven adenocarcinoma of the stomach without distant metastases (M0) and without infiltration of adjacent structures and organs.

3.1.2. D2 lymphadenectomy (based on Japanese gastric cancer guideline) 3.1.3. Age > 18 years 3.1.4. surgical resectability 3.1.5. follow-up time of at least 36 months.

Exclusion Criteria:

3.2.1. distant metastases (cM+) or infiltration of adjacent structures or organs (cT4b) and all primarily not resectable stages 3.2.2. Other types of lymphadenectomy lower than D2 3.2.3. Siewert type I and II Cardia cancers 3.2.2. Relapsed gastric cancers 3.2.3. malignant secondary disease, dated back < 5 years (exception: In-situ-carcinoma of the cervix uteri, adequately treated skin basal cell carcinoma)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4.1.1. This is a nationwide Multicenter observational retrospective study with matched comparison of two therapeutic strategies (NAC vs upfront surgery). Participating centers should have a hospital volume of at least 20 gastric resections for stomach cancer per year. We will include a) patients with cT>2, every cN, or b) patients with every T and N+, histologically proven adenocarcinoma of the stomach without distant metastases (M0) and without involvement of adjacent structures/organs, submitted either to pre- or peri-operative treatment and D2 gastrectomy or to upfront D2 gastrectomy, between January 2012 and December 2019, followed by adjuvant treatment when recommended. All patients who meet the inclusion/exclusion criteria will be registered into the study and classified to one of the two arms based on their treatment (a. Patients who underwent pre- or perioperative treatment and D2 gastrectomy - NAC or b. Patients submitted to upfront D2 gastrectomy- S).
Sampling Method: Probability Sample
Enrollment: 684 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3- and 5- year follow-up

SECONDARY OUTCOMES:
disease free survival (DFS) | [ Time Frame: 2-year follow-up ]
Perioperative Morbidity and Mortality | Time Frame: up to 2 months after surgery
R0-Resection rate | 2 months after surgery
Rate of NAC patients submitted to surgery | 3 years
Rate of NAC patients completing postoperative treatment | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- San Luigi University Hospital, Orbassano, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: Undecided